CLINICAL TRIAL: NCT06919133
Title: The Effect of Digital Markers in the Self-management of Depressive Symptoms - The MENTINA Randomized Controlled Parallel Group Trial
Brief Title: The Effect of Digital Markers in the Self-management of Depressive Symptoms
Acronym: MENTINA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); Research Centre of the German Foundation for Depression and Suicide Prevention (Unknown); Monsenso (Industry); Monsenso A/S as sponsor (Unknown)
Responsible Party: Principal Investigator, Lars Vedel Kessing, Professor, MD, Dr.Med., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101080651
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Mental Distress
Keywords: Depression; Mental distress; Smartphone; Trial; self-management
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-based self-monitoring and rule-based feedback (Experimental): The smartphone-based MENTINA app for daily self-monitoring of depressive symptoms and other symptoms + rule-based feedback based on self-monitoried data and sensor data from smartphones
  Interventions: Device: The MENTINA app
- Control (Placebo Comparator): The app is installed for outcome measures, but no access to the content of the app is provided.
  Interventions: Other: Control

INTERVENTIONS:
Device: The MENTINA app — A smartphone-based app is developed and used in this trial. The smartphone-based MENTINA app allows for daily self-monitoring of depressive symptoms such as mood, sleep, activity etc and rule-based feedback based on self-monitored data as well as collected sensor data. Libary with relevant content will also be available and incoorporated in the rule-based feedback.
  Arms: Smartphone-based self-monitoring and rule-based feedback
Other: Control — The MENTINA app is installed but no content and self-monitoring is available. No rule-based feedback. Only outcome measures can be done.
  Arms: Control

SUMMARY:
The purpose of the MENTINA trial is to investigate the effect of using the smartphone-based MENTINA app for self-monitoring of depressive symptoms and rule-based feedback in individuals with current or previous depression, psychological vulnerability, and increased risk of depression in a randomized controlled trial (RCT) over a 12-month trial period. The aim is to potentially offer the MENTINA app as a self-management tool for individuals with psychological vulnerability and/or depressive symptoms or episodes.

Method and Design:

International, multicenter (three centers), parallel-group, RCT. The active group is assigned the smartphone-based MENTINA app including rule-based data feedback. The control group uses the MENTINA app for questionnaire-based data collection (outcomes) and collection of sensor-based data.

Study Procedures:

The trial will be open-label and unblinded. The trial uses the self-reported Patient Health Questionnaire-9 score (PHQ-9) as the primary outcome measure. Scoring will take place every 14 days over the 12-month trial period. Depressive symptoms during the first 6 months of app use will also be evaluated as secondary outcomes.

Participants, Including Inclusion and Exclusion Criteria A total of 220 individuals will be included from each center (Denmark, Germany, and Spain) with psychological vulnerability (depressive symptoms and possibly previous depressive episodes). A total sample size of 660 participants will be included.

Inclusion criteria:

* Age 18 years or older
* Depressive symptoms, assessed by PHQ-9 > 8, AND/OR
* Current or previous depressive episode(s) (ICD-10 F32, F33)
* Owns and uses a smartphone
* Signed informed consent to participate

Exclusion criteria:

* ICD-10 diagnosis of dementia, schizophrenia, mania, or bipolar disorder, as well as ongoing substance abuse
* Current psychotic depression
* Current suicide risk
* Acute somatic illness requiring treatment (intensive care)
* Insufficient language skills in Danish, German or Spanish (depending on site)

Side Effects, Risks, and Disadvantages

Side effects and risks:

We do not expect any serious side effects from using the MENTINA app. Possible side effects could include increased focus on one's own illness, potentially worsening depressive symptoms and suicidal thoughts.

Recruitment of Participants The study population will consist of adults vulnerable to mental health issues, defined by a PHQ-9 score > 8 or previous depressive symptoms at the time of inclusion. Each study site will be responsible for local recruitment and follow-up.

DETAILED DESCRIPTION:
The intervention in the MENTINA trial consist of a smartphone app, which allows for daily monitoirng of symptoms such as mood, sleep, activity etc. Also, a library with content concerning depressive symptoms will be available.

Rules for feedback based of self-reported measures will be developed. Based on the self-reported measures participants will be suggested to read items from the library or call emergency health care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Depressive symptoms, assessed by PHQ-9 > 8, AND/OR
* Current or previous depressive episode(s) (ICD-10 F32, F33)
* Owns and uses a smartphone
* Signed informed consent to participate

Exclusion Criteria:

* ICD-10 diagnosis of dementia, schizophrenia, mania, or bipolar disorder, as well as ongoing substance abuse
* Current psychotic depression
* Current suicide risk
* Acute somatic illness requiring treatment (intensive care)
* Insufficient language skills in Danish, German or Spanish and english (depending on site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 items (PHQ-9) | From enrollment and during the study period of 12 months
  Differences between the intervention group and the control group in the total Patient Health Questionnaire 9 items (PHQ-9) score performed every 14th day during the 12-months trial period.

SECONDARY OUTCOMES:
Quality of Life | From enrollmetn to end of treatment af 12 months
  Differences between the intervention group and the control group in the level of quality of life according to the WHO Quality of life BREF16 (WHO QoL)
Generalized Anxiety Disorder 7 items scale (GAD-7) | From enrollment to end of treatment at 12 months
  Differences between the intervention group and the control group in the level of anxiety symptoms according to the Generalized Anxiety Disorder scale (GAD-7)
PHQ-9 | From baseline and during the 12 months study period
  * Monthly change in PHQ-9 scores
  * Response rate defined as the proportion of participants with ≥50% reduction in PHQ-9
  * Remission rate defined as PHQ-9 ≤9 and ≥5-point improvement
  * PHQ-9 scores at 6 months
  * Area Under the Curve (AUC) for PHQ-9 over the trial period
  * Subgroup analysis: differences between the two groups in PHQ-9 analyzed separately for:
    * People with mental distress (without lifetime depression)
    * People with a lifetime diagnosis of depression
Perceived Stress Scale (PSS) | From baseline and during the 12 months study period
  Differences between the group
User-reported healthcare contacts | From baseline and during the 12 months study period
  Number of healthcare contact during the study
Negative effects: Negative Effects Questionnaire (NEQ) | Form baseline and during the 12 months study period
  Differences between the two groups
PHQ-9 | From baseline and during the 12 months study period
  * Number of depressive episodes (based on PHQ-9)
  * Duration
  * Number of depression-free days (based on PHQ-9)

OTHER OUTCOMES:
Usability of the app: System Usability Scale (SUS) | From baseline and during the study period
  Usability of the app: System Usability Scale (SUS)
Perceived usefulness for patient-clinician communication | From baseline and during the trial period
  Qualitative interviews
Interviews with participants and clinicians/psychotherapists | From baseline and during the trial period
  Qualitative interviews on an subsample

CONTACTS AND LOCATIONS:
Locations (3):
- Psychiatric Center Copenhagen, Frederiksberg, Denmark
- Frankfurt University Hospital, Frankfurt, Germany
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Sensitive data that cannot be anonymised completely.

REFERENCES:
- [Derived] Faurholt-Jepsen M, Dyreholt MS, Kyster NB, Iversen N, Kortsen EM, Amann BL, Hogg B, Gatto D, Cordoba C, Petrovic M, Allenhof C, Schnitzspahn K, Reich H, Budtz-Jorgensen E, Kessing LV, Hegerl U. Effect of digital intervention in the self-management of depressive symptoms: the MENTINA trial - a study protocol for a randomised controlled parallel-group trial. BMJ Open. 2026 Feb 4;16(2):e115773. doi: 10.1136/bmjopen-2025-115773. PMID 41638726